CLINICAL TRIAL: NCT03653624
Title: Collection of Fully Anonymised Blood Pressure Data From Patients Undergoing Elective High Risk Surgery
Brief Title: Collection of Anonymised Blood Pressure Data During High Risk Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Directed Systems Limited (Industry)
Collaborators: University Hospital Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: BPA-DEP-001
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2018-08

CONDITIONS: Perioperative Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention is involved int his study. Fully anonymised blood pressure data will be collected from the vital signs monitors in the operating room.

SUMMARY:
This is a single centre, prospective, non-randomised clinical investigation to be undertaken at the Queen Elizabeth Hospital, Edgbaston, Birmingham.

The clinical investigation will collect fully anonymised perioperative blood pressure data from patients undergoing elective high risk surgery.

The Sponsor of this clinical investigation, Directed Systems Limited, is developing a new medical device, BP Assist, which provides guidance to anaesthetists in relation to the real-time management of patient cardiovascular physiology.

DETAILED DESCRIPTION:
This clinical investigation is designed to collect fully anonymised perioperative blood pressure data from patients undergoing high risk surgical procedures.

It is increasingly being recognised that in high risk surgery, the perioperative incidence and duration of hypotensive episodes (MAP <60mmHg) can adversely impact postoperative outcome.

Collecting continuous perioperative blood pressure data will enable hypotensive episodes to be recorded. Such data will be used to aid the development and testing of algorithms involved in generating the guidance provided by BP Assist.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older; undergoiing elective high risk surgery

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective high risk surgery at Queen Elizabeth Hospital, Birmingham, UK.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood pressure | Duration of each patient's surgery, up to 6 hours.
  The primary objective of this clinical investigation is to collect fully anonymised, continuous, perioperative blood pressure data from ten patients undergoing elective high-risk surgery. Systolic and mean arterial pressures will be recorded.

IPD SHARING:
Plan to Share IPD: No